CLINICAL TRIAL: NCT00041171
Title: Phase III Randomized Study of Hypericum Perforatum (St. John's Wort) Combined With Docetaxel in Patients With Unresectable Solid Tumors
Brief Title: Docetaxel and St. John's Wort in Treating Patients With Solid Tumors That Cannot Be Removed By Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was not activated.
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CALGB-60002; CDR0000069449 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Adult Solid Tumor; Breast Cancer; Head and Neck Cancer; Kidney and Urinary Cancer; Male Reproductive Cancer; Thorax and Respiratory Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; recurrent non-small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; stage III bladder cancer; recurrent bladder cancer; stage IV bladder cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; unspecified adult solid tumor, protocol specific; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage III squamous cell carcinoma of the lip and oral cavity; stage III basal cell carcinoma of the lip; stage III verrucous carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III inverting papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV inverting papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverting papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Urinary Bladder Neoplasms; Prostatic Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — Hypericum extract LI 160; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Arm 1: placebo + docetaxel (Experimental): Patients receive oral placebo three times daily on days 1-14 and docetaxel IV over 1 hour on day 15.
  Treatment in both groups repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Patients are followed for new primaries and survival only.
  Interventions: Drug: docetaxel; Other: placebo
- Arm 2: Hypericum perforatum + docetaxel (Experimental): Patients receive oral Hypericum perforatum three times daily on days 1-14 and docetaxel as in arm 1.
  Treatment in both groups repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Patients are followed for new primaries and survival only.
  Interventions: Drug: Hypericum perforatum; Drug: docetaxel
- Arm 3: Hypericum perforatum + docetaxel (Experimental): Patients receive docetaxel as in arm 1 and continue to receive their chronic regimen of Hypericum perforatum except on day 15.
  Treatment in both groups repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Patients are followed for new primaries and survival only.
  Interventions: Drug: Hypericum perforatum; Drug: docetaxel

INTERVENTIONS:
Drug: Hypericum perforatum
  Arms: Arm 2: Hypericum perforatum + docetaxel; Arm 3: Hypericum perforatum + docetaxel
Drug: docetaxel
Other: placebo
  Arms: Arm 1: placebo + docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. St. John's wort may interfere with the effectiveness of chemotherapy. It is not yet known if chemotherapy is more effective with or without St. John's Wort in treating solid tumors.

PURPOSE: Randomized phase III trial to compare the effectiveness of docetaxel with or without St. John's wort in treating patients who have solid tumors that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of Hypericum perforatum (St. John's Wort) on the pharmacokinetic clearance of docetaxel in patients with unresectable solid tumors.
* Determine the effect of Hypericum perforatum on the production and plasma concentrations of M4-C13-hydroxydocetaxel in these patients.
* Determine the effects of this drug on the pharmacodynamics of docetaxel in these patients.
* Determine the relationship between the effects of this drug on docetaxel metabolic clearance and CYP3A4/CYP3A5 genotype in these patients.
* Determine the relationship between the effect of this drug on docetaxel metabolic clearance and p-glycoprotein genotype in these patients.
* Determine the relationship between the effect of this drug on docetaxel clearance and pregnane receptor genotype in these patients.
* Assess compliance with this drug in these patients.
* Assess the steady state concentrations of hyperforin, one of the putative psychoactive components of Hypericum perforatum, in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients who have not been receiving chronic Hypericum perforatum (St. John's Wort) are assigned to group A, while a cohort of 8 patients who have been receiving chronic Hypericum perforatum are assigned to group B.

* Patients are randomized to 1 of 2 treatment arms.
* Arm I: Patients receive oral placebo three times daily on days 1-14 and docetaxel IV over 1 hour on day 15.
* Arm II: Patients receive oral Hypericum perforatum three times daily on days 1-14 and docetaxel as in arm I.
* Group B (non-randomized group): Patients receive docetaxel as in arm I and continue to receive their chronic regimen of Hypericum perforatum except on day 15.

Treatment in both groups repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed for new primaries and survival only.

PROJECTED ACCRUAL: Approximately 92 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unresectable solid tumor, including, but not limited to, the following:
* Lung cancer
* Breast cancer
* Head and neck cancer
* Bladder cancer
* Prostate cancer
* Must be suitable for treatment with single-agent docetaxel
* Hormone receptor status:
* Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* CTC 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than upper limit of normal (ULN)
* Alkaline phosphatase less than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN
* BUN no greater than 1.5 times ULN

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior bone marrow transplantation
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No prior docetaxel
* No more than 2 prior chemotherapy regimens
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal agents except steroids for adrenal failure or hormones for non-disease-related conditions (e.g., insulin for diabetes)

Radiotherapy:

* At least 3 weeks since prior radiotherapy
* No concurrent palliative radiotherapy

Surgery:

* At least 4 weeks since prior major surgery

Other:

* At least 6 months since prior Hypericum perforatum (St. John's Wort)
* At least 1 week since prior CYP3A enzyme inducers including:
* Phenobarbital
* Phenytoin
* Carbamazepine
* Lamotrigine
* Rifampin
* Rifabutin
* Isoniazid
* Sulfinpyrazone
* Pioglitazone
* Anti-HIV drugs such as efavirenz or nevirapine
* At least 1 week since prior CYP3A enzyme inhibitors including:
* Erythromycin
* Clarithromycin
* Azithromycin
* Roxithromycin
* Ketoconazole
* Fluconazole
* Itraconazole
* Metronidazole
* Chloramphenicol
* Ritonavir
* Saquinavir
* Indinavir
* Nelfinavir mesylate
* Delavirdine
* Amiodarone
* Cyclosporine
* Tacrolimus
* Sirolimus
* Nefazodone
* Fluvoxamine
* No concurrent CYP3A enzyme inducers
* No concurrent CYP3A enzyme inhibitors
* No ethanol (especially red wine), grape fruit juice, or seville orange juice (CYP3A enzyme inhibitor) within 3 days before or after receiving docetaxel

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lionel D. Lewis, MD, Study Chair — Norris Cotton Cancer Center